CLINICAL TRIAL: NCT04848051
Title: Implementing Fit Kit Colorectal Cancer (CRC) Screening in High Risk Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2000030006; 2P30CA016359-39 (NIH)
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer
Keywords: Health Screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CRC screening reminder (Experimental): Participants randomized to the CRC Reminder arm will receive reminder that they are due/overdue for CRC screening
  Interventions: Behavioral: CRC screening reminder
- CRC Reminder & Short message (Experimental): Participants randomized to the CRC Reminder & short message arm will receive reminder that they are due/overdue for CRC screening and short message to encourage screening
  Interventions: Behavioral: CRC Reminder & Short message
- CRC Reminder and Navigation Program (Experimental): Participants randomized to the CRC reminder and navigation program arm will receive reminder that they are due/overdue for CRC screening and short message to participate in the health navigation program that will connect participants to individually tailored resources and assistance
  Interventions: Behavioral: CRC Reminder and Navigation Program
- CRC Reminder & CRC education (Experimental): Participants randomized to the CRC reminder and CRC education program arm will receive reminder that they are due/overdue for CRC screening and offered short educational program conducted online
  Interventions: Behavioral: CRC Reminder & CRC education

INTERVENTIONS:
Behavioral: CRC screening reminder — Participants randomized to the CRC Reminder arm will receive reminder that they are due/overdue for CRC screening
  Arms: CRC screening reminder
Behavioral: CRC Reminder & Short message — Participants randomized to the CRC Reminder & short message arm will receive reminder that they are due/overdue for CRC screening and short message to encourage screening
  Arms: CRC Reminder & Short message
Behavioral: CRC Reminder and Navigation Program — Participants randomized to the CRC reminder and navigation program arm will receive reminder that they are due/overdue for CRC screening and short message to participate in the health navigation program that will connect participants to individually tailored resources and assistance
  Arms: CRC Reminder and Navigation Program
Behavioral: CRC Reminder & CRC education — Participants randomized to the CRC reminder and CRC education program arm will receive reminder that they are due/overdue for CRC screening and offered short educational program conducted online
  Arms: CRC Reminder & CRC education

SUMMARY:
The purpose of this study is to understand best strategies for engaging high risk populations in a primary care setting to improved adherence to colorectal cancer screening guidelines. The results will be used to identify best practices that are scalable to other high-risk populations who are due or overdue for colorectal cancer (CRC) screening.

DETAILED DESCRIPTION:
This is a prospective implementation science study that will test 4 different approaches to increase colorectal cancer screening in a local primary care setting that provides services to individuals who are under-resourced. The interventions will include reminders from primary care providers with and without additional information and/or services to help complete colorectal cancer screening. A review of electronic medical records will be used to identify baseline information assessing risk factors and personal and family CRC history. For arm 3 of the study, participants may elect to enroll in our existing health navigation program. If so, additional baseline information will be collected, including information on Social Determinants of Health (SDOH). For arm 4 of the study, a questionnaire will be used to assess knowledge about colorectal cancer screening. The questionnaire will be repeated after the intervention (informational video). For all arms of the study, the primary outcome (engagement on CRC screening, receipt of CRC screening, results of CRC screening) will be collected through EPIC.

ELIGIBILITY:
Inclusion Criteria:

* be 50-74 years of old at the time of enrollment
* have one valid medical encounter with CSHHC Columbus Ave. location or Dixwell location between the dates of 11/01/2019 and 11/30/2020

Exclusion Criteria:

• Documented history of colorectal cancer

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3127 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Total number of participants who completed their colorectal cancer screening | 18 months
  The total number of participants that completed their colorectal cancer screening will be measured between the different arms

SECONDARY OUTCOMES:
Time to engagement | 18 months
  The time to engagement will be measured as the days between reminder or reminder + intervention and days to screening among the 4 arms
Screening outcomes: results of screening | 18 months
  Screening outcomes will be defined as the following: descriptive summaries of the result of screening among the 4 arms.
Screening outcomes: follow up | 18 months
  Screening outcomes will be defined as the following: descriptive summaries of need and completion of follow up among the 4 arms.
Screening outcomes: biopsy results | 18 months
  Screening outcomes will be defined as the following: descriptive summaries of biopsy results (if needed) among the 4 arms.
Screening outcomes: diagnostic results | 18 months
  Screening outcomes will be defined as the following: descriptive summaries of the diagnostic result(s) among the 4 arms.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Jones, Principal Investigator — Yale University
Locations (1):
- Cornell Scott Hill Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided